CLINICAL TRIAL: NCT03074045
Title: Multi-center, Randomized, Open-label, Parallel-group Study to Evaluate User Satisfaction With and Tolerability of the Low-dose Levonorgestrel (LNG) Intrauterine Delivery System (IUS) With 16 μg LNG/Day Initial in Vitro Release Rate (LCS16) in Comparison to a Combined Oral Contraceptive (COC) Containing 30 μg Ethinyl Estradiol and 3 mg Drospirenone (Yarina®) in Young Nulliparous and Parous Women (18 - 29 Years) Over 12 Months of Use (With an Option for Extended Use of LCS16 for up to 5 Years)
Brief Title: LCS16 vs. COC User Satisfaction and Tolerability Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17878
Record Dates: First submitted 2017-03-03; First posted 2017-03-08 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Contraception
Keywords: Intrauterine; Birth control
MeSH Terms: interventions — Levonorgestrel; Ethinyl Estradiol; drospirenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (Experimental): LCS16 (Low-dose LNG IUS)
  Interventions: Drug: Levonorgestrel (Kyleena, BAY86-5028)
- Reference (Active Comparator): COC (Yarina)
  Interventions: Drug: Ethinyl estradiol and drospirenone (Yarina, BAY86-5131)

INTERVENTIONS:
Drug: Levonorgestrel (Kyleena, BAY86-5028) — Low-dose LNG IUS with an initial in vitro release rate of 16 μg LNG/day, used continuously. The total LNG content in LCS16 is 19.5 mg. Administered intrauterine, for 12 months with an option for extended use for up to 5 years
  Arms: Test
Drug: Ethinyl estradiol and drospirenone (Yarina, BAY86-5131) — COC tablet containing 30 μg ethinyl estradiol and 3 mg drospirenone (taken on cycle days 1-21, inclusive, followed by a 7-day tablet-free week) for 12 months
  Arms: Reference

SUMMARY:
To evaluate user satisfaction in young nulliparous and parous women (18-29 years of age [inclusive]), using LCS16 compared to a COC over a period of 12 months.

ELIGIBILITY:
Inclusion Criteria:

* The subject has signed and dated the Informed Consent Form (ICF).
* The subject is healthy when requesting contraception.
* The subject is between 18 - 29 years of age (inclusive) at the time of signing the ICF.
* The subject has normal or clinically insignificant cervical smear for oncocytology (i.e. Pap test) not requiring further follow up (a cervical smear has to be taken at the Screening Visit [Visit 1] or a normal result has to have been documented within the previous 6 months).
* The subject has a history of regular (i.e., endogenous cyclicity without hormonal contraceptive use) cyclic menstrual periods (length of cycle 21 - 35 days), as confirmed by the subject.
* The subject is willing and able to attend the scheduled study visits and to comply with the study procedures.

Exclusion Criteria:

* Pregnancy or current lactation (less than 6 weeks postpartum or since abortion before the Screening Visit)
* Infected abortion or postpartum endometritis within 3 months prior to the Screening Visit.
* Chronic, daily use of drugs that may increase serum potassium levels.
* Undiagnosed abnormal genital bleeding.
* Acute cervicitis or vaginitis (until successfully treated).
* Lower urinary tract infection (until successfully treated).
* Acute or recurrent pelvic inflammatory disease or conditions associated with increased risk for pelvic infections.
* Congenital or acquired uterine anomaly including fibroids, in the opinion of the investigator, which would interfere with insertion and/or retention of the intrauterine system (i.e., if they distort the uterine cavity).
* Cervical neoplasia, uterine or cervical malignancy, or sex hormone-dependent tumors.
* History of migraine, focal migraine with asymmetrical visual loss or other symptoms indicating transient cerebral ischemia.

Ages: 18 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 145 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2018-09-03 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Overall satisfaction rate | 12 months
  5-point Likert item
  1. Very satisfied
  2. Satisfied
  3. Neither satisfied nor dissatisfied
  4. Dissatisfied
  5. Very dissatisfied

SECONDARY OUTCOMES:
Number of adverse events | Up to 5 years
  at 1, 6 and 12 months for all subjects during the comparative part of the study.
  at the end of Year 2, Year 3, Year 4 and Year 5 only for subjects, who elect to enter the LCS16 extension phase.
Discontinuation rates | Up to 5 years
  at 1, 6 and 12 months for all subjects during the comparative part of the study.
  at the end of Year 2, Year 3, Year 4 and Year 5 only for subjects, who elect to enter the LCS16 extension phase.
Bleeding pattern | Up to 12 months
  Only during the comparative part of the study
User satisfaction and bleeding questionnaire | Up to 12 months
  At 6 and 12 months after the start of study treatment (or at early termination for those subjects discontinuing the study before completion of the 12 months) for all subjects during the comparative part of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (9):
- Russia (9):
  - Altai State Medical University, Barnaul
  - Scientific Center of family health & human reprod. problems, Irkutsk
  - Krasnoyarsk State Medical University, Krasnoyarsk
  - City Clinical Hospital #13 Moscow, Moscow
  - LLC Reafan, Novosibirsk
  - Medical Center "Avicenna", Novosibirsk
  - LLC Medical center PRIME ROSE, Saint Petersburg
  - Smolensk State Medical University, Smolensk
  - Regional perinatal center, Yaroslavl

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

REFERENCES:
- [Result] Suturina L.V., Dikke G.B. Experience in the use of low-dosed levonorgestrelcontaining intrauterine system Kyleena LNG and combined oral contraceptive containing 30 mcg ethinyl estradiol and 3 mg drospirenone in young women. Akusherstvo i Ginekologiya/Obstetrics and Gynecology. 2021; 11: 230-236 (in Russian)